CLINICAL TRIAL: NCT00169468
Title: Phase II Study of the Association of Velcade to R-CHOP in the Treatment of B Cell Lymphoma
Brief Title: Association of Velcade to R-CHOP in the Treatment of B Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Collaborators: Association pour le Développement de la Recherche Clinique et Informatique en Onco-Hématologie (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-CHOP VELCADE
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: B Cell Lymphoma
Keywords: B Lymphoma; Velcade; Chemotherapy
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Bortezomib

INTERVENTIONS:
Drug: Rituximab -CHOP plus Velcade

SUMMARY:
The primary objective of this study is to evaluate the response rate and toxicity of the association R-CHOP with two schedules of administration of Velcade, in B-cell CD 20 + lymphoma patients, aged from 18 to 80 years

The goal is to get a response rate at least at what observed with R-CHOP alone and will be evaluates with a sequential test.

The other objective is to evaluate the toxicity

DETAILED DESCRIPTION:
The association of the monoclonal antibody Rituximab to chemotherapy regimen of B-cell lymphoma is associated with an increase response rate and event free survival when compared to chemotherapy alone (Coiffier et al NEJM 2002). It has been observed in almost all histological type of B-cell lymphomas. No significant increase of toxicity was observed especially in the most used regimen CHOP and the association R-CHOP is a standard for most B-cell malignancies CD20 positive.

However, in patients with diffuse large cell lymphoma progress should be made as the complete response rate is below 75% in most situation and in low grade lymphoma, although patients respond well to chemotherapy complete remission rate averaged generally 50% (Marcus et al 2003), Czuczman et al 1999) .

There is a need to improve this association with new innovative agent. Before running randomized study it is important to evaluate the like hood of getting improvement by phase 2 study testing tolerance and efficacy on a well established regimen.

Bortezomib (Velcade formerly PS 341) is a proteasome inhibitor which has shown promising activity in the treatment of refractory myeloma. As single agent in indolent lymphomas, administered twice per weeks for 2 weeks followed by one week rest period it has already showed activity in phase 2 study. It is well tolerated and main toxicity was neuropathy and thrombocytopenia.

Proteasome inhibitors can act through multiple mechanisms to arrest tumor growth, tumor spread, and angiogenesis. In vitro studies have shown a synergistic effect of the association of Velcade and doxorubicin on myeloma cell lines resistant to chemotherapy.

Association of Velcade to standard chemotherapy regimen is under study with the aim of improving on the results.

Association of Velcade to one of the most efficient treatment of B-cell lymphoma, R-CHOP, might increase the response rate.

However, different schedules should be explored in order to better appreciate efficacy and toxicity.

This randomized phase 2 study is designed to evaluate the response rate and the toxicity of two schedules of administration of Velcade in association with R-CHOP. The aim of the study is to establish a well tolerated regimen giving a response rate in the limit upper/lower of what is observed with conventional R-CHOP used in all the different histological subtypes of B cell lymphomas patients requiring treatment.

The heterogeneity of the population will preclude any meaningful subgroup analysis.

It is important to evaluate tolerability before exploring the efficacy of this new regimen in large randomized studies or in specific phases II study which will need 50 patients for each subgroup of patients.

ELIGIBILITY:
Inclusion Criteria:

• Patients with one of the following B-cell Lymphoma CD 20 positive : Mantle cell, Marginal zone, lymphocytic, follicular requiring treatment, Histological transformation from low grade to high grade, diffuse large cell without adverse prognostic factors defined by the international prognostic index (IPI)

* Aged from 18 to 80 years
* Untreated with chemotherapy except with Chlorambucil or Cyclophosphamide per os alone less than 6 months
* Previous radiotherapy except if localized
* Performance status < 3
* Signed inform consent

Exclusion Criteria:

* Other type of lymphomas: Burkitt, T cell, CD 20 negative
* Central nervous system or meningeal involvement
* Contraindication to any drug contained in the chemotherapy regimen
* HIV disease, active hepatitis B or C
* Treatment with polychemotherapy before except with Chlorambucil or Cyclophosphamide per os less than 6 months
* Prior extended radiotherapy
* Any serious active disease or co-morbid medical condition (according to investigator's decision )
* Renal deficiency (clearance < 30 ml/mn), liver deficiency (bilirubin > 30 mmol/l) unless related to lymphoma
* Neuropathy> grade 2 within 14 days before enrollment
* Platelets < 30.109/l within 14 days before enrollment
* Neutrophils < 1.0 109/l within 14 days before enrollment
* Women with pregnancy or without adequate method of contraception
* Any history of active cancer during the last two years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Rate of complete remission | 1 year
Number of SAE | 1 year

SECONDARY OUTCOMES:
Duration of response | 1 year
Progression free survival | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: christian Gisselbrecht, MD PHD, Principal Investigator — Lymphoma Study Association
Locations (4):
- France (4):
  - Hôpital Saint-Louis, Paris, Paris 10
  - Institut Gustave Roussy, Villejuif, Villejuif Cedex
  - Hôpital Henri Mondor, Créteil
  - Hôpital Lyon Sud, Pierre-Bénite

REFERENCES:
- [Background] Czuczman MS, Grillo-Lopez AJ, White CA, Saleh M, Gordon L, LoBuglio AF, Jonas C, Klippenstein D, Dallaire B, Varns C. Treatment of patients with low-grade B-cell lymphoma with the combination of chimeric anti-CD20 monoclonal antibody and CHOP chemotherapy. J Clin Oncol. 1999 Jan;17(1):268-76. doi: 10.1200/JCO.1999.17.1.268. PMID 10458242
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Background] 44. Marcus R, et al. (2003). An International Multi-Centre, Randomized, Open-Label, Phase III Trial Comparing Rituximab Added to CVP Chemotherapy to CVP Chemotherapy Alone in Untreated Stage III/IV Follicular Non-Hodgkins Lymphoma. Blood, 102, issue 11, (abstract 87).
- [Background] O'Connor O, Wright J, Moskowitz CH, Muzzy J, MacGregor-Cortelli B, Hamlin P, Straus D, Trehu E, Schenkein DP, Zelenetz AD. Promising activity of the proteasome inhibitor bortezomib (VELCADE) in the treatment of indolent non-Hodgkin's lymphoma and mantle cell lymphoma: ASH poster session 517-II. J Natl Compr Canc Netw. 2004 Nov;2 Suppl 4:S21-2. PMID 19791425